CLINICAL TRIAL: NCT05768555
Title: Investigation of the Effects of Single Session Whole Body Vibration Training Applied with Different Frequencies in Hypertensive Patients
Brief Title: Whole Body Vibration Training Applied with Different Frequencies in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Bilge Köksal, Master of Science, Dokuz Eylul University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DokuzEU-HT-001
Record Dates: First submitted 2023-02-23; First posted 2023-03-14 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: hypertension; whole body vibration
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Whole body vibration intervention at 40 Hz (Active Comparator): 40 Hz frequency WBVT
  Interventions: Other: Whole body vibration intervention at 40 Hz
- Whole body vibration intervention at 25 Hz (Active Comparator): 25 Hz frequency WBVT
  Interventions: Other: Whole body vibration intervention at 25 Hz
- Whole body vibration intervention at 0 Hz (Active Comparator): 0 Hz frequency WBVT
  Interventions: Other: Whole body vibration intervention at 0 Hz

INTERVENTIONS:
Other: Whole body vibration intervention at 40 Hz — Whole body vibration intervention will be performed with the Power Plate Pro 5 device (Power Plate International, London, UK). Whole body vibration training will be performed at a frequency of 40 Hz. Individuals will perform; static squat, dynamic toe raise, static abduction and dynamic squat exercises in both hips on a vibrating platform. All exercises will consist of 45 seconds of vibration and 15 seconds of rest. Each exercise will be repeated three times. Total intervention time will be 15 minutes.
  Arms: Whole body vibration intervention at 40 Hz
Other: Whole body vibration intervention at 25 Hz — Whole body vibration intervention will be performed with the Power Plate Pro 5 device (Power Plate International, London, UK). Whole body vibration training will be performed at a frequency of 25 Hz. Individuals will perform; static squat, dynamic toe raise, static abduction and dynamic squat exercises in both hips on a vibrating platform. All exercises will consist of 45 seconds of vibration and 15 seconds of rest. Each exercise will be repeated three times. Total intervention time will be 15 minutes.
  Arms: Whole body vibration intervention at 25 Hz
Other: Whole body vibration intervention at 0 Hz — Whole body vibration intervention will be performed with the Power Plate Pro 5 device (Power Plate International, London, UK). Whole body vibration training will be performed at a frequency of 0 Hz. Individuals will perform; static squat, dynamic toe raise, static abduction and dynamic squat exercises in both hips on a vibrating platform. All exercises will consist of 45 seconds of vibration and 15 seconds of rest. Each exercise will be repeated three times. Total intervention time will be 15 minutes.
  Arms: Whole body vibration intervention at 0 Hz

SUMMARY:
At least 36 volunteers with a diagnosis of hypertension in the Department of Cardiology of Dokuz Eylul University and who meet the criteria for follow-up and inclusion will participate in the study. The aim of this study is to compare the acute effects on atherosclerosis, heart rate variability, blood pressure, perceived exertion, energy expenditure, and muscle strength of using different frequencies in whole body vibration training (WBVT) in hypertensive patients. Individuals will perform; static squat, dynamic toe raise, static abduction and dynamic squat exercises in both hips on a vibrating platform. In each session, a different frequency (0,25 and 40 Hz) will be applied. 0 Hz, 25 Hz and 40 Hz sessions will be randomized to last 15 minutes. Demographic and clinical information of the participants will be questioned.Before and after the sessions; hemodynamic and pulmonary responses, vascular responses, heart rate variability and quadriceps femoris muscle strength will be measured. In addition, energy expenditure will be recorded during the sessions.

DETAILED DESCRIPTION:
Hypertension is one of the most common chronic diseases and it is an important global public health problem. In cardiac rehabilitation programs, aerobic exercise, resistance exercise and a combination of aerobic and resistance exercise are recommended to reduce cardiovascular risk. Whole body vibration training has also started to be used among new applications in the cardiac rehabilitation programs. Whole body vibration training has been reported as an effective and safe approach for both healthy and cardiovascular diseased women and men. It has been shown to be beneficial in improving atherosclerosis and blood pressure in hypertensive patients. In whole body vibration training, frequencies of 20-40 Hz are generally used for hypertensive elderly patients. However, the optimal frequency in this population has not been fully determined. For these reasons, the aim of the study is to compare the acute effects of using different frequencies in whole body vibration training in hypertensive patients.

Whole body vibration intervention will be performed with the Power Plate Pro 5 device (Power Plate International, London, UK). Whole body vibration training will be performed at three different frequencies (0, 25 and 40 Hz). Each patient will complete the training in these 3 frequencies in random order and on different days. Before and after the sessions; hemodynamic and pulmonary responses, vascular responses, heart rate variability and quadriceps femoris muscle strength will be measured. In addition, energy expenditure will be recorded during the sessions.Individuals will perform; static squat, dynamic toe raise, static abduction and dynamic squat exercises in both hips on a vibrating platform. All exercises will consist of 45 seconds of vibration and 15 seconds of rest. Each exercise will be repeated three times. Total intervention time will be 15 minutes. Participants will perform whole body vibration trainings at different frequencies in a randomized order with at least one day apart.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with hypertension
* Being clinically stable
* Becoming a volunteer
* Walking independently
* Not taking medication or hormone therapy in the year before the study
* Lack of regular exercise habit (<60 minutes/week of exercise)

Exclusion Criteria:

* Having a serious cardiovascular/pulmonary condition
* Having an operation in the last 6 months
* Presence of acute thrombosis
* Presence of arrhythmia
* Presence of unstable angina
* Recent decompensated heart failure
* Recent myocardial infarction
* Using an assistive device to walk
* Neurological disorders (such as stroke, Parkinson's)
* Being diagnosed with vertigo
* Being diagnosed with epilepsy
* Kidney failure and history of kidney stones
* Hip or knee implants
* Recent fractures or injuries (<6 months).
* Using a prosthesis
* Pregnancy
* Participation in any training program in the 3 months before study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | Change from the baseline to the first minutes after the intervention
  Arterial stiffness will be measured with a noninvasive method with the help of the SphygmocorXCEL device, which can automatically measure with the cuff. The patient's age(years), gender(male), blood pressure(mmHg), height(cm), weight(kg), carotid-sternal notch distance between the artery, carotid-femoral artery as the distance between the entered data to the computer after increasing pressure over the brachial artery through a transducer (augmentation index) and again, carotid-femoral pulse wave velocity via the artery (pulse wave velocity) measurements will be made.
Heart rate variability | Change from the baseline to the first minutes after the intervention
  Heart rate variability will be assessed by heart rate variability (HRV), a non-invasive measurement. Sympathetic and parasympathetic autonomic function will be evaluated with HRV software. HRV provides time and frequency domain parameters associated with autonomic function.
Blood pressure | Change from the baseline to the first minutes after the intervention
  Systolic and diastolic blood pressure will be measured with a sphygmomanometer.

SECONDARY OUTCOMES:
Muscle strength | Change from the baseline to the first minutes after the intervention
  Lower extremity quadriceps muscle strength will be evaluated with a digital dynamometer (Lafayette, USA). The knee and hip joint will be measured in a 90-degree sitting position. The dynamometer will be stabilized by a plastic sheath and an inelastic belt. Measurements will be performed on both lower extremities and for each extremity, the best value will be recorded from the measurements repeated 3 times. Higher values indicate better quadriceps muscle strength.
Energy expenditure | During exercise intervention, average 15 minutes
  Energy expenditure during whole body vibration trainings with different frequencies will be evaluated using the activity monitor. The activity monitor will be attached to the upper arm.
Heart rate | Change from the baseline to the first minutes after the intervention
  Heart rate will be recorded with Polar heart rate monitor.
Perceived effort | Change from the baseline to the first minutes after the intervention
  The degree of perceived effort will be evaluated with the Modified Borg scale(M.Borg 0-10). As the modified borg score of the person increases, the perceived effort will increase.
Respiratory frequency | Change from the baseline to the first minutes after the intervention
  It will be counted manually for 30 seconds and multiplied by two.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Savcı, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No